CLINICAL TRIAL: NCT05185245
Title: Liver Transplantation for Non-Resectable Colorectal Liver Metastasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LITORALE2020
Record Dates: First submitted 2021-12-10; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-04

CONDITIONS: Liver Metastasis Colon Cancer; Colorectal Cancer
Keywords: liver transplantation; non-resectable colorectal liver metastasis
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver Transplantation (Experimental)
  Interventions: Procedure: Liver Transplantation

INTERVENTIONS:
Procedure: Liver Transplantation — Liver Transplantation for Non-Resectable Colorectal Liver Metastasis

SUMMARY:
The study aims to evaluate the efficacy of liver transplantation in the context of non-resectable colorectal liver metastasis. The primary endpoint is the overall survival in this group of patients while the secondary endpoint is the disease-free survival.

Patients included in this protocol will be evaluated either for whole or partial liver transplantation from deceased or living donors.

Type of different transplantations proposed are as follows:

1. Whole liver graft or partial liver (split) from a deceased donor
2. Partial liver graft retrieved from a deceased donor and orthotopically implanted after having performed a left hepatectomy in the recipient.
3. Partial liver graft retrieved from a deceased donor and heterotopically implanted if total hepatectomy can not be performed.
4. Partial liver graft retrieved from a living donor and orthotopically implanted after having performed total hepatectomy.
5. Partial liver graft retrieved from a living donor and orthotopically implanted after having after having performed a left hepatectomy in the recipient.
6. Partial liver graft retrieved from a living donor and heterotopically implanted if total hepatectomy can not be performed.

In cases 2-3-5-6 total hepatectomy of native liver can be secondarily performed after having achieved a proper graft hypertrophy in order to avoid a small for size syndrome

ELIGIBILITY:
Inclusion Criteria:

* Primary tumor resected according to standard oncological practice, p≤T4a, R0 resection
* Colorectal liver metastasis considered as non-resectable either up-front or after previous hepatic resections
* No local recurrence of primary colon cancer confirmed by Positron Emission Tomography, Computed Tomography and colonoscopy
* No extra-hepatic metastatic disease confirmed by Positron Emission Tomography and Computed Tomography
* Good performance status Eastern Cooperative Oncology Group 0 or 1
* Neutrophils > 1.000
* Patients who received at least one line of chemotherapy for at least 3 months with partial response or stable disease according to modified Response Evaluation Criteria in Solid Tumours
* Carcino-Embryonic Antigen < 80 µg/L or reduction of ≥ 50% of highest Carcino-Embryonic Antigen level observed
* Written informed consent
* No other contraindications to liver transplantation

Exclusion Criteria:

* Presence of other malignancies
* Local recurrence of primary tumor
* Extra-hepatic metastatic disease
* Patients who did not receive any neoadjuvant or adjuvant therapy
* Palliative resection of primary tumor
* Any other reason, according to the investigators, that could be a contraindication to protocol enrollment

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5 years

SECONDARY OUTCOMES:
Disease-Free Survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Italy